CLINICAL TRIAL: NCT03799445
Title: Phase 2 Study (With Safety Lead in) of the Safety, Tolerability and Efficacy of Anti-CTLA4 (Ipilimumab) and Anti-PD-1 (Nivolumab) in Combination With Radiation Therapy to 50-66 Gy in Low-Intermediate Volume, Local-Regionally Advanced HPV-Positive Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Brief Title: Ipilimumab, Nivolumab, and Radiation Therapy in Treating Patients With HPV Positive Advanced Oropharyngeal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0381; NCI-2018-03260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0381 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-13; First posted 2019-01-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Human Papillomavirus Positive Oropharyngeal Squamous Cell Carcinoma; Oropharyngeal Basaloid Carcinoma; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Posterior Tongue Squamous Cell Carcinoma; Soft Palate Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IVA Oropharyngeal Squamous Cell Carcinoma AJCC v7; Tonsillar Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab, IMRT) (Experimental): Patients receive nivolumab IV over 30 minutes on days 1, 15, and 29 and ipilimumab IV over 30 minutes on day 1. Treatment repeats every for 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of cycle 2, patients also undergo IMRT 5 days a week (Monday-Friday) for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Biological: Ipilimumab; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the side effects and best dose of ipilimumab, nivolumab, and radiation therapy and how well they work in treating patients with advanced human papillomavirus (HPV) positive oropharyngeal squamous cell carcinoma. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving ipilimumab, nivolumab, and radiation therapy may work better in treating patients with HPV positive oropharyngeal squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety, tolerability and feasibility of ipilimumab and nivolumab when administered concurrently with reduced-field radiotherapy (intensity-modulated radiation therapy [IMRT]).

II. To evaluate the clinical complete response rate to ipilimumab, nivolumab and IMRT with reduced field at six months as indicated by fluorodeoxyglucose - positron emission tomography/computed tomography (FDG-PET/CT) post completion of radiation therapy (RT).

III. To evaluate the 2-year progression-free survival (PFS) rate of subjects with low-intermediate volume, local-regionally advanced, human papilloma virus (HPV)-positive squamous cell carcinoma of the head and neck (SCCHN) treated with ipilimumab, nivolumab and reduced-field IMRT.

SECONDARY OBJECTIVES:

I. To evaluate overall response rate to six weeks of induction immunotherapy (IO).

II. To evaluate the frequency of pharyngeal dysphasia as measured by Dynamic Imaging (Dynamic Imaging Grade of Swallowing Toxicity [DIGEST]) grade on modified barium swallow (MBS) and patient-reported symptoms (MD Anderson Dysphagia Inventory [MDADI]) at 6 month, 1 and 2 years after radiotherapy ([IMRT].

III. To measure acute and chronic toxicities per Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (CTCAE PRO).

IV. To measure acute toxicity profiles at the end of radiation therapy and IO and at 6 months.

V. To measure late toxicity profiles at 1 and 2 years. VI. To determine local and regional control at 6 and 12 months. VII. To determine patterns of failure (local-regional relapse vs. distant) at 1 and 2 years.

VIII. To determine overall survival (OS) at 1 and 2 years.

CORRELATIVE OBJECTIVES:

I. To evaluate associations between total mutational load, interferon (INF) gamma score, T cell clonality at diagnosis with clinical response to induction, combination CTLA-4 PD-1 checkpoint blockade.

II. To evaluate changes in the tumor immune microenvironment (CD8 + INF gamma score, T cell clonality, in tumor biopsy specimens pre and post induction immunotherapy (IO).

III. To evaluate dynamic changes in and clearance of oral HPV and cell-free deoxyribonucleic acid (cfDNA) viral load during therapy and to investigate associations with PFS and OS.

EXPLORATORY OBJECTIVES:

I. To evaluate changes in peripheral blood lymphocyte phenotypes and serum cytokine profiles before and after induction IO.

II. To evaluate changes in the T cell receptor repertoire in tumor-infiltrating lymphocyte (TIL) and the peripheral blood in tumor biopsy specimens pre and post induction IO.

III. To determine the negative and positive predictive values (NPV and PPV) of FDG-PET/CT 12-14 weeks after end of RT for 1 year and 2 year PFS and OS.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on days 1, 15, and 29 and ipilimumab IV over 30 minutes on day 1. Treatment repeats every for 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of cycle 2, patients also undergo IMRT 5 days a week (Monday-Friday) for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically newly confirmed diagnosis of squamous cell carcinoma (including the histological variants of papillary or basaloid) of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls)
* Clinical American Joint Committee on Cancer (AJCC) 7th edition stage T1N2a-N2CM0, T2N1-N2CM0, T3N0-N2CM0, equivalent to AJCC 8th edition stage 1 and 2 (T1 N2, T2 N1-N2, T3 N0-N2) excluding T1N0-N1 and T2N0 (Brian O'Sullivan et al. 2016)
* Tumor positive for p16 immunohistochemistry (IHC) (defined as greater than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells) and HPV DNA in situ hybridization or HPV messenger ribonucleic acid (mRNA) RNAScope. Repeat samples may be required if adequate diagnostic tissue is unavailable for testing
* Zubrod Performance Status of 0-1
* Patients must have radiographically evident measurable disease at the primary site or at nodal stations per response evaluation criteria in solid tumors (Response Evaluation Criteria in Solid Tumors [RECIST]) 1.1 documented by diagnostic quality CT or magnetic resonance imaging (MRI) of the neck with contrast within 28 days prior to registration; a FDG-PET/CT of the neck performed for the purposes of radiation planning is acceptable as a substitute if the CT is of diagnostic quality
* Diagnostic quality cross sectional imaging of the thorax within 28 days prior to registration. A 18-FDG-PET/CT or conventional CT are acceptable
* FDG-PET/CT of the neck is required within 28 days prior to registration for comparison to post treatment FDG-PET/CT. Note: Repeat imaging for variability within 96 hours of this time frame should be allowed to avoid unnecessary re-imaging and its financial and potential physical consequences for patients
* History and physical exam within 1 month prior to registration
* Fiberoptic exam with laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) by radiation oncologist, medical oncologist or ear, nose, throat (ENT)/head and neck surgeons within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 2 weeks prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 2 weeks prior to registration)
* Hemoglobin >= 8.0 g/dl (within 2 weeks prior to registration); Note: The use of transfusion or other intervention to achieve Hgb >= 8.0 g/dl is acceptable
* Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) >= 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula (within 2 weeks prior to registration)
* Bilirubin < 2 mg/dl (within 2 weeks prior to registration)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the upper limit of normal (within 2 weeks prior to registration)
* Sodium (Na), potassium (K), chloride (Cl), glucose, calcium (Ca), magnesium (Mg), albumin, amylase, lipase, thyroid stimulating hormone (TSH) within 2 weeks prior to registration
* Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential
* Seronegative for active hepatitis-B or hepatitis-C infection and seronegative for human immunodeficiency virus (HIV)
* Mandatory submission of hematoxylin and eosin (H&E) and paraffin-embedded tumor block or unstained slides

Exclusion Criteria:

* Cancers of the oral cavity (oral tongue, floor mouth, alveolar ridge, buccal or lip), or the nasopharynx, hypopharynx, or larynx, even if p16 positive
* Carcinoma of the neck of unknown primary site origin (even if p16 positive)
* Definitive clinical or radiologic evidence of metastatic disease or adenopathy below the clavicles
* Gross total excision of both primary and nodal disease with curative intent; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease
* Simultaneous primary cancers or separate bilateral primary tumor sites
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable; patients who have received PD-1/PD-L1 or CTLA4 therapy for a previous malignancy are not eligible
* Prior RT to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity defined as any of the following: Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration; hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; a diagnosis of immunodeficiency or use of any form of systemic immunosuppressive therapy. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Steroid premedications for contrast allergy allowed
* Has evidence of active, non-infectious pneumonitis
* Has received a live vaccine within 30 days of planned start of study therapy
* Pregnancy or breast-feeding; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* History of severe hypersensitivity or contraindication to CT or PET contrast material uncontrolled with pre-medications (steroids, antihistamines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) (safety lead-in) | Up to 28 days post-completion of radiation therapy
  Defined as any >= grade 3 adverse event (Common Terminology Criteria for Adverse Events [CTCAE], version [v.] 4) that is related to immunotherapy (IO) that does not resolve to grade 1 or less within 28 days.
Complete response rate (Phase II) | At 6 months
Progression-free survival (PFS) (Phase II) | From start of therapy to progression or disease or death from any cause, assessed up to 2 years

SECONDARY OUTCOMES:
Number of patients who experience a >= grade 3 treatment-related adverse event (safety lead-in) | Up to 28 days post-completion of radiation therapy
Number of patients who tolerated protocol therapy (safety lead-in) | Up to 12 weeks (end of cycle 2)
  The number of patients who tolerated protocol therapy, including completion of radiotherapy without a treatment break and who were administered immunotherapy (IO) will be assessed.
Number of patients who achieve a clinical complete response (safety lead-in) | Up to 28 weeks after radiation therapy
Incidence of acute and chronic adverse events (Phase II) | Up to 3 months from the end of intensity-modulated radiation therapy (IMRT)
  Incidence of adverse events (acute and chronic toxicities) will be assessed per CTCAE Patient Reported Outcome (PRO).
Acute toxicity profiles (Phase II) | At the end of radiation therapy, end of IO, and 6 months
  Will be assessed by CTCAE v 4.
Number of patients who experience >= grade 3 treatment-related adverse event (Phase II) | At the end of radiation therapy, end of IO, and 6 months
Late toxicity profiles (Phase II) | At 1 and 2 years
  Will be assessed per CTCAE v 4.
Patient-reported swallowing outcomes (Phase II) | At 1 and 2 years
Patterns of failure (local-regional relapse versus [vs] distant) (Phase II) | At 1 and 2 years
Overall survival (Phase II) | At 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org